CLINICAL TRIAL: NCT01555554
Title: Effect of Prophylactic, Perioperative Propranolol on Peri- and Postoperative Complications in Patients With Post Traumatic Stress Disorder
Brief Title: Perioperative Propranolol in Patients With Post Traumatic Stress Disorder (PTSD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to meet enrollment goals.
Sponsor: University of California, San Francisco (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Northern California Institute of Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: W81XWH-10-2-0078
Record Dates: First submitted 2012-03-05; First posted 2012-03-15 (Estimated); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Post-traumatic stress disorder; Propranolol; surgery; anesthesia
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Propranolol; propranolol CR

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol Hydrochloride (Experimental)
  Interventions: Drug: Propranolol Hydrochloride
- Placebo Group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Propranolol Hydrochloride — Propranolol will be taken for a total of 14 days. On the morning of the surgery, prior to entry into the operating room, patients will receive the first dose of the study drug (the PDR recommended starting dose of Propranolol XL- Extended Release). Patients will take one 60 mg pill on the morning of surgery.
  On post operative day #1, patients will take one pill of receive propranolol XL 80 mg (once daily by mouth).
  On post operative days #2-#9, patients will take one pill of propranolol XL 120 mg (once daily by mouth).
  On post operative days #10-11, patients will take one pill of propranolol XL 80 mg (once daily by mouth).
  On post operative days #12-13, patients will take one pill of propranolol XL 60 mg (once daily by mouth).
  This will complete the course of propranolol.
  Other Names: Inderal; Inderal LA; Avlocardyl; Avlocardyl Retard; Deralin; Dociton; Inderalici; InnoPran XL; Sumial; Anaprilinum; Bedranol SR Sandoz
  Arms: Propranolol Hydrochloride
Other: Placebo — The placebo pill will be taken for a total of 14 days. On the morning of the surgery, prior to entry into the operating room, patients will receive the first placebo pill to be taken once daily by mouth.
  On post operative days #1-13, patients will take one placebo pill (once daily by mouth).
  This will complete the course of the placebo.
  Arms: Placebo Group

SUMMARY:
Understanding what treatments may facilitate perioperative care of Veterans with posttraumatic stress disorder (PTSD) is of great importance to the U.S. health care system.

Patients with PTSD are characterized by elevated central nervous system catecholamine concentrations and exaggerated and prolonged adrenergic responses to stress stimuli. At present, there are no data on the effects of perioperative beta blocker therapy in patients with PTSD, despite the rising significance of PTSD in Veteran populations.

This prospective, double-blind study proposes to randomize 150 Veterans with PTSD scheduled for orthopedic, thoracic or vascular surgery at the San Francisco VA Medical Center to either a 14-day course of propranolol or placebo. This study will then follow these Veterans for a one-year period to evaluate the effects of the intervention on Veterans' surgical outcomes.

The investigators hypothesize that patients with PTSD randomized to the propranolol group will demonstrate a reduced incidence of perioperative and postoperative morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects scheduled for any surgical procedure under general anesthesia or combined general-regional anesthesia, with the exception of open-heart or intracranial surgery. Regional anesthesia includes: 1) Epidural anesthesia, 2) Sub-arachnoid block (spinal), or 3)any regional nerve block
2. Anticipated postoperative hospital admission (defined as at least one overnight hospital stay)

Exclusion Criteria:

Veterans will be excluded if:

1. They are on beta blocker therapy at the time of the preoperative baseline assessment
2. They report sensitivity or allergies to propranolol, or a history of PTSD exacerbation with prior propranolol therapy
3. Veterans who fulfill the AHA/ACC level I recommendation criteria for perioperative beta blocker therapy (e.g., metoprolol, atenolol) and should not be randomized to placebo group
4. Medical exclusions criteria: high grade heart block without pacemaker (all patients with 2nd and 3rd degree heart block), marked resting bradycardia (heart rate ≤ 55 beats per minute), blood pressure < 100 mmHg, uncompensated congested heart failure, severe hyperactive airway disease, and Raynaud's disease
5. Pregnancy
6. Current use of medication that may involve potentially dangerous interaction with propranolol
7. Circumstances that, in the opinion of the principal investigator, would preclude participation in a study of this type (e.g. medical concerns or difficulty in long-term followup).
8. Open-heart surgery and intracranial surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-05; Primary Completion 2018-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
ICU length of stay | Truncated at 30 days after admission to ICU
  Measured using patient medical records
Hospital length of stay | Truncated at 30 days after admission to ICU
  Measured using patient medical records
Postoperative delirium | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Measured using Confusion Assessment Method (CAM-CAM-ICU)
Postoperative renal dysfunction | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Measured using Serum Creatinine laboratory values

SECONDARY OUTCOMES:
Perioperative complications | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Measured using patient medical records
Pain intensity | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using the Numerical Rating Scale
Pain unpleasantness | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using the Numerical Rating Scale
Analgesics use | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using patient medical records
Length of intubation and mechanical ventilation | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Measured using patient medical records
Post Traumatic Stress Disorder symptomatology | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using the Posttraumatic Diagnostic Scale (PDS)
Quality of Life | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using Short Form-36 Questionnaire (SF-36)
Functional status | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using Short Form-36 Questionnaire (SF-36)
Sleep Quality | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using the Pittsburgh Sleep Quality Index (PSQI)
Depression symptoms | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using the Beck Depression Inventory (BDI)
Postoperative Neurocognitive Dysfunction Score | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using the Mini Mental State Examination (MMSE)
30-day, 3-month, and 1-year mortality | Participants will be followed from preoperative baseline to 1 year postoperative
  Measured using patient medical records
Postoperative complications | Participants will be followed to 1 year postoperative
  Measured using patient medical records

CONTACTS AND LOCATIONS:
Overall Officials: Marek Brzezinski, M.D., Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States